CLINICAL TRIAL: NCT05305742
Title: Evaluation of Postoperative Pain and Bacterial Load Reduction After Canal Preparation With ProTaper Ultimate Versus ProTaper Gold Rotary Systems in Patients With Necrotic Maxillary Premolars (Randomized Clinical Trial)
Brief Title: Evaluation of Postoperative Pain and Bacterial Load Reduction With ProTaper Ultimate Versus ProTaper Gold Rotary Systems
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Khaled Hassan Abed, Dentist / Master Degree Student at Faulty of Dentistry, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ENDO3-3-5
Record Dates: First submitted 2021-12-24; First posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Protaper Ultimate (Experimental)
  Interventions: Other: Instrument Design
- Protaper Gold (Active Comparator)
  Interventions: Other: Instrument Design

INTERVENTIONS:
Other: Instrument Design — Research the effect of different instrument designs on root canal preparation by evaluating bacterial count reduction and post-operative pain

SUMMARY:
This study aims to research the effect of different instrument designs by comparing protaper ultimate versus protaper gold systems on root canal preparation by evaluating bacterial count reduction and post-operative pain following single visit treatment in patients with necrotic pulp in maxillary premolar teeth.

ELIGIBILITY:
Inclusion Criteria:

* Patient's age ranges between 22 to 45 years with no sex predilection.
* Medically free patients.
* Maxillary permanent premolar teeth:

  * Diagnosed clinically with pulp necrosis.
  * Absence of pain.
  * Radiographic evidence of two roots or single root with double canals.
  * Slight widening in the periodontal membrane space or with peri-apical radiolucency
  * No response to cold pulp tester and ethyl chloride spray.
* Patients who can understand Modified Visual Analogue Scale (VAS).
* Patients' acceptance to participate in the trial.

Exclusion Criteria:

* Medically compromised patients.
* Pregnant women.
* If analgesics or antibiotics have been administrated by the patient during the past 24 hours preoperatively.
* Patients reporting bruxism or clenching.
* Teeth with:

  i. Vital teeth. ii. Single canal maxillary premolar teeth iii. Association with swelling or fistulous tract. iv. Acute peri-apical abscess and swelling. v. Mobility Grade II or III. vi. Pocket depth more than 5mm. vii. Previous root canal therapy. viii. Non-restorable teeth: Hopeless tooth
* Immature teeth.
* Radiographic evidence of external or internal root resorption vertical root fracture, perforation, calcification, root caries.

Ages: 22 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
Post Operative Pain | Postoperative pain will be measured by modified Visual Analogue Scale immediately after the end of treatment, and at 6, 12, 24 and 48 hours.
  Intensity of pain felt after endodontic treatment recorded by the patient using modified Visual Analogue Scale where 0=no pain, 1-3=mild pain, 4-6=moderate pain and 7-10=severe pain

SECONDARY OUTCOMES:
Number of needed analgesic tablets in case of intolerable pain | Patient will be contacted after 48 hours after endodontic treatment to know the number of analgesic tablets taken
  The patient will record the number of analgesic tablets taken in case of intolerable pain
Antibacterial Effectiveness | First as a Baseline (T0): After the access cavity Sample 1 will be taken, after 15 minutes (T1) mechanical instrumentation will be done and Sample 2 will be taken, after 5 minutes from T1 (T2) final irrigation will be done and Sample 3 will be taken.
  Bacterial counting using agar Culture technique